CLINICAL TRIAL: NCT06590896
Title: A Phase 2, Multicenter Open-Label Extension Study to Evaluate the Long-term Safety of Cenobamate in Japanese Subjects With Partial Onset Seizures
Brief Title: Safety of Cenobamate in Japanese Subjects With Partial Onset Seizures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-2017-02; jRCT2031220198 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-08-08; First posted 2024-09-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Cenobamate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cenobamate (Experimental)
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — Cenobamate will be orally administered once daily.

SUMMARY:
To evaluate the long-term safety and tolerability of cenobamate in Japanese epilepsy patients with partial seizures

ELIGIBILITY:
Inclusion Criteria:

* Subjects completed Study YKP3089C035 by SK Life Science.

Exclusion Criteria:

* Subjects that have previously discontinued for any reason from the Core study (YKP3089C035).
* Any significant changes to the medical history of the subject that in the opinion of the investigator, could affect the safety of the subject.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidences of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, an average of 4 years
  The incidences of adverse events (AEs) and serious adverse events (SAEs) will be recorded.
Urinalysis(pH) | Through study completion, an average of 4 years
  Measurement of urine pH.
Urinalysis(Specific Gravity) | Through study completion, an average of 4 years
  Measurement of urine specific gravity (g/mL).
Urinalysis(Protein) | Through study completion, an average of 4 years
  Measurement of urine protein (mg/dL).
Urinalysis(Glucose) | Through study completion, an average of 4 years
  Measurement of urine glucose (mg/dL).
Urinalysis(Ketone) | Through study completion, an average of 4 years
  Measurement of urine ketone (mg/dL).
Urinalysis(Bilirubin) | Through study completion, an average of 4 years
  Measurement of urine bilirubin (mg/dL).
Urinalysis(Blood) | Through study completion, an average of 4 years
  Measurement of urine blood (presence/absence).
Urinalysis(Nitrite) | Through study completion, an average of 4 years
  Measurement of urine nitrite (presence/absence).
Urinalysis(Urobilinogen) | Through study completion, an average of 4 years
  Measurement of urine urobilinogen (mg/dL).
Urinalysis( Microscopic Examination) | Through study completion, an average of 4 years
  Microscopic examination of urine (if abnormal).
Liver function tests(total protein) | Through study completion, an average of 4 years
  Measurement of total protein(g/dL)
Liver function tests(albumin) | Through study completion, an average of 4 years
  Measurement of albumin(g/dL)
Liver function tests(total bilirubin) | Through study completion, an average of 4 years
  Measurement of total bilirubin(mg/dL)
Liver function tests(aspartate transaminase) | Through study completion, an average of 4 years
  Measurement of aspartate transaminase(U/L)
Liver function tests(alanine aminotransferase) | Through study completion, an average of 4 years
  Measurement of alanine aminotransferase(U/L)
Liver function tests(alkaline phosphatase) | Through study completion, an average of 4 years
  alkaline phosphatase(U/L)
Liver function tests(gamma-glutamyl transferase) | Through study completion, an average of 4 years
  Measurement of gamma-glutamyl transferase(U/L)
Hematology(Hemoglobin) | Through study completion, an average of 4 years
  Measurement of hemoglobin(g/dL)
Hematology(hematocrit) | Through study completion, an average of 4 years
  Measurement of hematocrit(%)
Hematology(white blood cell count) | Through study completion, an average of 4 years
  Measurement of white blood cell count（/μL）
Hematology(red blood cell count) | Through study completion, an average of 4 years
  Measurement of red blood cell count（/μL)
Hematology(mean corpuscular volume) | Through study completion, an average of 4 years
  Measurement of mean corpuscular volume(fL)
Hematology(mean corpuscular hemoglobin) | Through study completion, an average of 4 years
  Measurement of mean corpuscular hemoglobin(pg)
Hematology(red blood cell distribution width) | Through study completion, an average of 4 years
  Measurement of red blood cell distribution width(％)
Hematology(platelet count) | Through study completion, an average of 4 years
  Measurement of platelet count(/μL)
Serum chemistry(blood urea nitrogen) | Through study completion, an average of 4 years
  Measurement of blood urea nitrogen(mg/dL)
Serum chemistry(calcium) | Through study completion, an average of 4 years
  Measurement of calcium(mg/dL)
Serum chemistry(chloride) | Through study completion, an average of 4 years
  Measurement of chloride(mEq/L)
Serum chemistry(creatinine) | Through study completion, an average of 4 years
  Measurement of creatinine(mg/dL)
Serum chemistry(total bilirubin) | Through study completion, an average of 4 years
  Measurement of total bilirubin(mg/dL)
Serum chemistry(direct bilirubin) | Through study completion, an average of 4 years
  Measurement of direct bilirubin(mg/dL)
Serum chemistry(alkaline phosphatase) | Through study completion, an average of 4 years
  Measurement of alkaline phosphatas（U/L）
Serum chemistry(alanine aminotransferase) | Through study completion, an average of 4 years
  Measurement of alanine aminotransferase(U/L)
Serum chemistry(gamma-glutamyl transferase) | Through study completion, an average of 4 years
  Measurement of gamma-glutamyl transferase(U/L)
Serum chemistry(total protein) | Through study completion, an average of 4 years
  Measurement of total protein(g/dL)
Serum chemistry(albumin) | Through study completion, an average of 4 years
  Measurement of albumin(g/dL)
Serum chemistry(globulin) | Through study completion, an average of 4 years
  Measurement of globulin(g/dL)
Serum chemistry(sodium) | Through study completion, an average of 4 years
  Measurement of sodium(mEq/L)
Serum chemistry(potassium) | Through study completion, an average of 4 years
  Measurement of potassium(mEq/L)
Serum chemistry(phosphorus) | Through study completion, an average of 4 years
  Measurement of phosphorus(mq/dL)
Serum chemistry(glucose) | Through study completion, an average of 4 years
  Measurement of glucose(mq/dL)
Heart rate | Through study completion, an average of 4 years
  heart rate (beats per minute)
Respiratory Rate | Through study completion, an average of 4 years
  Respiratory Rate (breaths per minute),
Blood Pressure | Through study completion, an average of 4 years
  blood pressure, both of systolic and diastolic (mm Hg)
Electrocardiogram (ECG) Findings | Through study completion, an average of 4 years
  ECG findings, including heart rate (beats per minute), PR Interval (milliseconds), PQ Interval (milliseconds), RR Interval (milliseconds), QRS Interval (milliseconds), and QT Interval (milliseconds), will be recorded.
Columbia-Suicide Severity Rating Scale (C-SSRS) Scores | Through study completion, an average of 4 years
  Scores on the Columbia-Suicide Severity Rating Scale (C-SSRS) will be recorded. Questions regarding suicide are recorded as yes or no, and the percentage of subject with suicide risk (yes) is assessed.

SECONDARY OUTCOMES:
Percentage Change in all partial seizure frequency per 28-Day | Through study completion, an average of 4 years
  It will confirm the frequency of partial seizures at 28-day intervals and calculate the percentage change until the study is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (29):
- Japan (29):
  - Ehime University Hospital, Ehime
  - Department of Neurology and Stroke Center, Southern Tohoku Clinic., Fukushima
  - Hiroshima University Hospital, Hiroshima
  - NHO Kure Medical Center and Chugoku Cancer Center, Hiroshima
  - Asahikawa Medical University Hospital, Hokkaido
  - Itami City Hospital, Hyōgo
  - JA-Ibaraki Tsuchiura Kyodo General Hospital, Ibaraki
  - University of Tsukuba Hospital, Ibaraki
  - Kagoshima University Hospital, Kagoshima
  - Tanaka Neurosurgical Clinic, Kagoshima
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Yokohama City University Hospital, Kanagawa
  - Kumamoto Ezuko Rehabilitation Medical Center, Kumamoto
  - NHO Nagasaki Medical Center, Nagasaki
  - Koide Clinic of Epilepsy and Neurological Disorders, Osaka
  - Osaka University Hospital, Osaka
  - Shintokukai Nii Neurosurgery and Psychiatry Clinic, Osaka
  - Ochiai Brain Clinic, Saitama
  - TMG ASAKA Medical Center, Saitama
  - Sakurai Clinic, Shiga
  - NHO Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka
  - Seirei Hamamatsu General Hospital, Shizuoka
  - Seirei Mikatahara General Hospital, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Medical Hospital, Tokyo Medical and Dental University, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - NHO Yamagata National Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No